CLINICAL TRIAL: NCT07035236
Title: Clinical, Radiographic and Histologic Evaluation of Tenting the Schneiderian Membrane Using Titanium Mesh for Maxillary Sinus Lift Procedure: A Randomized Controlled Study
Brief Title: Evaluation of Tenting the Schneiderian Membrane of the Maxillary Sinus Using Titanium Mesh.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Hedra sherif, Freelance dentist, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 967/2025
Record Dates: First submitted 2025-06-05; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Maxillary Sinus Floor Augmentation
Keywords: Tenting; Schneiderian membrane

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium mesh group (study group) (Experimental): Group I (study group) the Schneiderian membrane will be elevated using titanium mesh fixed by screws
  Interventions: Procedure: maxillary sinus lifting
- Screws group (control group) (Active Comparator): Group II (control group) will have stainless steel screws/pins placed bucco-palatally to maintain the elevated membrane and stabilize the formed blood clot
  Interventions: Procedure: Maxillary sinus lifting

INTERVENTIONS:
Procedure: maxillary sinus lifting — The schneiderian membrane will be tented using titanium mesh.
  Arms: Titanium mesh group (study group)
Procedure: Maxillary sinus lifting — The Schneiderian membrane will be elevated using bone screws
  Arms: Screws group (control group)

SUMMARY:
Twenty posterior maxillary edentulous sites requiring open sinus augmentation for staged dental implant placement will be studied. Group I (study group) the maxillary sinus membrane will be elevated using titanium mesh fixed by bone screws. Group II (control group) will have stainless steel screws/pins placed bucco-palatally to maintain the elevated membrane and stabilize the formed blood clot. Platelet rich fibrin (PRF) will be placed at the site of elevated membrane in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult male/female patients with age interval 18:60 years old.
* Patients with one or more teeth requiring implant supported dental restoration in atrophic maxilla.
* Alveolar bone height less than 5 mm at the defective site.
* Good oral hygiene.
* Patient's consensual agreement to be enrolled in the study.

Exclusion Criteria:

* Medically compromised patients with conditions contraindicating surgery (eg. uncontrolled diabetics, bisphosphonate intake, radio or chemotherapy).
* Patients with active infection at or related to the site of surgery (eg. acute sinusitis).
* Heavy smokers.
* Patients not indicated for an implant supported restoration at the time of enrollement (eg. active/untreated periodontal disease). (Patients developing any medical condition that interferes with the outcomes after enrolment in the study will be excluded).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Histological evaluation of gained bone quality | 6 months
  Using Hematoxin and Eosin stains
Radiographic Bone gain after maxillary sinus lift | 6 months
  Using Cone Beam CT

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT07035236/Prot_SAP_ICF_000.pdf